CLINICAL TRIAL: NCT01798186
Title: Pharmacokinetic and Pharmacodynamic Effects of Passive Cannabis Inhalation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NA_00082269
Record Dates: First submitted 2013-02-18; First posted 2013-02-25 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Cannabis Toxicology
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Between subjects Phase I study
Who Masked: Participant
Masking Description: Participants are blind to the THC concentrations of cannabis being administered
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cannabis 5% THC, No Ventilation (Experimental): Participants in this condition will be passively exposed to second-hand cannabis smoke from cannabis containing 5% THC and in a room with no ventilation.
  Interventions: Drug: Cannabis
- Cannabis 11% THC, No Ventilation (Experimental): Participants in this condition will be passively exposed to second-hand cannabis smoke from cannabis containing 11% THC and in a room with no ventilation.
  Interventions: Drug: Cannabis
- Cannabis 11% THC, Ventilation (Experimental): Participants in this condition will be passively exposed to second-hand cannabis smoke from cannabis containing 11% THC in a room with active ventilation.
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — Participants will be exposed to cannabis smoke present in ambient air
  Other Names: Marijuana

SUMMARY:
This primary aim of this study is to assess the effects of passive (second-hand) inhalation of cannabis smoke on toxicological analysis of "native" oral fluid (saliva), urine and blood specimens. The results of this study will help inform the validity of oral fluid as a biomarker of cannabis exposure and to determine whether, and for how long, passive inhalation of cannabis smoke could result in a positive toxicology result.

ELIGIBILITY:
Participants must:

* Be between the ages of 18 and 45
* Be in good general health based on a physical examination, medical history, vital signs, 12-lead ECG and screening urine and blood tests
* Demonstrate ability to expectorate 3-5 mL of "native" oral fluid over a 5-minute period
* Be willing and able to abstain from use of any over-the-counter (OTC) or prescription drugs (other than birth control medications) after providing written informed consent and continuing until discharged from the study. OTC antacids may be taken up to 12 hours prior to dosing
* Not be pregnant or nursing (if female), and using effective birth control. All females must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at clinic admission.
* Have a body mass index (BMI) in the range of 19 to 33 kg/m2
* Have head hair that is at least 4-6 cm (approximately two inches) in length on the back of the head.
* Blood pressure at Screening Visit must not exceed a systolic blood pressure (SBP) of 140 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
* Must not have history of significant medical or psychiatric illness judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
* Cannot have been enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing.
* No history of panic/anxiety reaction to extended periods of confinement in close quarters, smoke filled areas, or tight social situations.
* No history of adverse reactions to cannabis exposure, whether via direct use or passive exposure.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 3 experimental sessions. Additionally, participants were recruited to smoke cannabis in order to generate the smoke that was passively inhaled by the experimental groups.
Groups:
- Cannabis 5% THC, no Ventilation: passive exposure to 5% THC in an unventilated room
- Cannabis 11% THC, no Ventilation: passive exposure to 11% THC cannabis smoke in an unventilated room
- Cannabis 11% THC, Ventilated: passive exposure to 11% THC cannabis smoke in a room with active air ventilation
- Active Smokers: Participants that smoked cannabis
Period: Overall Study
Arm/Group | Cannabis 5% THC, no Ventilation | Cannabis 11% THC, no Ventilation | Cannabis 11% THC, Ventilated | Active Smokers
Started | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cannabis 5% THC, no Vent: passive exposure to 5% THC cannabis smoke, unventilated room
- Cannabis 11% THC, no Vent: passive exposure to 11% THC cannabis smoke, unventilated room
- Cannabis 11% THC, Vent: passive exposure to 11% THC cannabis smoke, ventilated room
- Smokers: cannabis smokers
- Total: Total of all reporting groups
Arm/Group | Cannabis 5% THC, no Vent | Cannabis 11% THC, no Vent | Cannabis 11% THC, Vent | Smokers | Total
Number analyzed (Participants) | 6 | 6 | 6 | 8 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (3) | 29 (9) | 30 (8) | 29 (6) | 28 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 3 | 12
  Male | 3 | 3 | 3 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 6 | 6 | 4 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 2 | 5
  White | 3 | 5 | 5 | 5 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Delta-9-tetrahydrocannabinol (THC) Cmax in Blood
Description: After exposure to cannabis, we will conduct a pharmacokinetic analysis of THC in blood collected.
Time Frame: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 22, 26, 30, and 34 hours post cannabis exposure
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 5% THC Cannabis, no Vent: passive exposure to 5%THC cannabis smoke in unventilated room
- 11% THC Cannabis Smoke, no Vent: passive exposure to 11% THC cannabis smoke in unventilated room
- 11% THC Cannabis, Vent: passive exposure to 11% THC cannabis smoke in ventilated room
Arm/Group | 5% THC Cannabis, no Vent | 11% THC Cannabis Smoke, no Vent | 11% THC Cannabis, Vent
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 1.4 (0.5) | 3.07 (1.6) | 0.5 (0.4)

2. Secondary Outcome: Delta-9-tetrahydrocannabinol (THC) Cmax in Oral Fluid
Description: After exposure to cannabis, we will conduct a pharmacokinetic analysis of THC in oral fluid.
Time Frame: Samples collected 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 22, 26, 30, and 34 hours post cannabis exposure
Measure: Mean (Full Range); unit: ng/mL
Groups:
- 5%THC Cannabis, no Ventilation: passive exposure to 5% THC cannabis smoke, no room ventilation
- 11%THC Cannabis, no Ventilation: passive exposure to 11% THC cannabis smoke, no room ventilation
- 11% THC Cannabis, no Ventilation: passive exposure to 5% THC cannabis smoke, with active room ventilation
Arm/Group | 5%THC Cannabis, no Ventilation | 11%THC Cannabis, no Ventilation | 11% THC Cannabis, no Ventilation
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 34 [5 to 86] | 82 [12 to 308] | 17 [2 to 75]

3. Secondary Outcome: Subjective VAS Drug Effect
Description: Visual analog scale (0-100; not at all to extremely) of subjective "Drug Effect"
Time Frame: immediately post cannabis exposure.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- 5%THC, no Vent: passive 5% THC cannabis smoke, no room ventilation
- 11% THC Cannabis, Ventilated: passive exposure to 11% THC cannabis smoke in ventilated room
Arm/Group | 5%THC, no Vent | 11% THC Cannabis Smoke, no Vent | 11% THC Cannabis, Ventilated
Number analyzed (Participants) | 6 | 6 | 6
mm | 6 (5) | 23 (13) | 3 (4)

ADVERSE EVENTS:
Time Frame: 2 days
Groups:
- 5% THC Cannabis Smoke, no Ventilation: passive exposure to 5%THC cannabis smoke in unventilated room
- 11% THC Cannabis Smoke, no Ventilation: passive exposure to 11%THC cannabis smoke in unventilated room
- 11% THC Cannabis Smoke, Ventilation: passive exposure to 11%THC cannabis smoke in ventilated room
Arm/Group | 5% THC Cannabis Smoke, no Ventilation | 11% THC Cannabis Smoke, no Ventilation | 11% THC Cannabis Smoke, Ventilation
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No